CLINICAL TRIAL: NCT05929677
Title: Linking Impulsivity Domains and Subjective Response to Alcohol in Young Adults Using Lab and Daily Assessment Methods
Brief Title: Impulsivity Domains and Subjective Response
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jessica Weafer (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Jessica Weafer, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 71127; R01AA029488 (NIH)
Record Dates: First submitted 2023-05-19; First posted 2023-07-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder
Keywords: Addiction; Alcohol; Young adult; Impulsivity; Prevention; Subjective response
MeSH Terms: conditions — Alcoholism; Behavior, Addictive; Impulsive Behavior | interventions — Sodium Chloride; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Alcohol, Then Placebo, then Free-access session (Experimental): participants will complete two intravenous administration sessions in the lab during which they will receive alcohol then placebo (saline), followed by a third lab session in which they will have free-access to self-administer alcohol (up to 120mg% BrAC) and placebo intravenously for 60 min
  Interventions: Drug: Placebo; Drug: Alcohol
- Placebo, Then Alcohol, then Free-access session (Experimental): participants will complete two intravenous administration sessions in the lab during which they will receive placebo (saline) then alcohol, followed by a third lab session in which they will have free-access to self-administer alcohol (up to 120mg% BrAC) and placebo intravenously for 60 min
  Interventions: Drug: Placebo; Drug: Alcohol

INTERVENTIONS:
Drug: Placebo — Participants receive placebo (saline) intravenously. They will also have the opportunity to self-administer saline during the 60-minute free-access IV self-administration period in session 3.
  Other Names: Saline
Drug: Alcohol — Participants receive alcohol intravenously, clamped at BrACs of 20mg%, 40mg%, and 60mg%. They will also have the opportunity to self-administer alcohol (up to 120mg% BrAC) during the 60-minute free-access IV self-administration period in session 3.

SUMMARY:
Findings from this project will determine the relationship between two vulnerability factors for Alcohol Use Disorder (AUD) in young adults: impulsivity and subjective response to alcohol. The results will identify badly needed, novel targets for prevention and treatment efforts to simultaneously reduce impulsivity and subjective responses in at-risk young adults.

DETAILED DESCRIPTION:
Young adult alcohol misuse is an urgent, growing public health crisis, as young adults have the highest alcohol use disorder rates of any age group with rates increasing in young women. Interventions for this population are hampered by small effects, few options and lack of tailoring to salient risk factors. A recent review in Addiction argued that research informing interventions fails to account for the complexity of relationships among factors contributing to young adult alcohol misuse. These needs will be addressed by examining relationships between two cardinal etiologic risk factors: impulsivity and subjective response to alcohol (SR). Despite theoretical and biological links between them, little is known about relations between the two risk factors, or how associations between them may promote young adult alcohol misuse longitudinally and on a momentary or daily basis. Prior theory and evidence linking impulsivity and positive, rewarding alcohol effects have been primarily learning and expectancy based. Here, based on exciting preliminary results, the researchers posit an inherent, biological link between impulsivity and high-risk SR (elevated stimulation and dampened sedation). This research is nascent with multiple gaps in knowledge. These gaps will be addressed by examining impulsivity pre-drinking, SR and alcohol use in a lab setting and via seven 10-day daily assessment periods over 2 years using ecological momentary assessment (EMA) (N=250, 50% female). Using self-report and both lab and mobile tasks, the investigators will characterize 3 unique, established impulsivity domains: poor inhibitory control, delay discounting and negative urgency. SR will be assessed at successive breath alcohol levels using precision intravenous (IV) methods in the lab, followed by opportunity to self-administer more IV alcohol. SR will also be measured at roughly comparable, estimated blood alcohol levels via daily EMA methods. This design enables testing of SR early in a drinking event as a predictor of in-lab and daily alcohol use, along with alcohol use and consequences over time, plus SR's potential role as a mediator of impulsivity/alcohol relations. Recent findings indicate daily changes in impulsivity predict subsequent drinking and consequences. These types of changes are challenging to capture with lab methods only. Daily measures also enable modeling of both person-level individual differences and daily, within-subject effects. However, there are no published studies relating daily impulsivity and SR measures. In this study, investigators will: 1) determine relations between lab-based impulsivity and SR; 2) determine relations between daily impulsivity and SR; and 3) relate impulsivity and SR to alcohol misuse longitudinally.

Researchers hypothesize impulsivity will relate to heightened stimulation and less sedation following alcohol and that SR will partially mediate relations between impulsivity and alcohol misuse. Evidence of links between specific impulsivity domains and SR longitudinally and on a momentary/daily basis will point to specific intervention targets to ameliorate two critical vulnerability factors for young adult alcohol misuse. Thus, investigators will: 1) identify mechanisms of alcohol action and 2) facilitate prevention and treatment research: two NIAAA priority areas.

Findings from this project will determine the relationship between two vulnerability factors for Alcohol Use Disorder (AUD) in young adults: impulsivity and subjective response to alcohol. The results will identify badly needed, novel targets for prevention and treatment efforts to simultaneously reduce impulsivity and subjective responses in at-risk young adults. As such, the project is directly relevant to NIAAA's mission to identify mechanisms of alcohol action and facilitate prevention and treatment research.

ELIGIBILITY:
Inclusion Criteria:

* 21-25 years old
* Report drinking to an estimated BAC > .08% at least once in the past 30 days based on responses on the Timeline Followback (TLFB)
* Report drinking at least twice weekly in the past 30 days based on responses on the TLFB
* Fluency in English

Exclusion Criteria:

* Any serious medical problems (e.g., liver disease, cardiac abnormality, pancreatitis, diabetes, neurological problems, and gastrointestinal disorders)
* Body weight < 110 or > 210 pounds
* Axis I psychiatric disorders including substance use disorder other than mild or moderate alcohol or mild cannabis use disorder
* Current alcohol withdrawal or history of medically-assisted detoxification
* Two positive breath alcohol concentration (BrAC) readings (i.e., > 0.00%) at an in-person screening appointment or experimental session
* Positive urine screen for illegal drugs other than cannabis
* Currently seeking or past-12-month history of inpatient or intensive treatment for addictive behaviors
* Current psychotropic medication use or receipt of a prescription for these medications in the past 30 days
* Psychosis or other psychiatric disability
* Pregnancy, nursing or lack of reliable birth control use for women
* Report smoking > 5 cigarettes per day (to avoid acute nicotine effects or withdrawal during experimental sessions)

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Lab Subjective Response to Alcohol (SR) | 70 minutes
  Participants provide subjective ratings of stimulation and sedation using the Brief Biphasic Alcohol Effects Scale (scores from 0 to 10 where a higher number means more stimulation/sedation).
Ecological Momentary Assessment (EMA) Subjective Response to Alcohol (SR) | 10 days
  Participants provide subjective ratings of stimulation and sedation using the Brief Biphasic Alcohol Effects Scale (scores from 0 to 10 where a higher number means more stimulation/sedation) using the EMA app.
Change in Breath Alcohol Concentration (BrAC) | 60 minutes
  Highest BrAC in mg% taken by breathalyzer during the free-access period
Number of alcohol drink units self administered | 60 minutes
  participants can self-administer alcohol infusions by pushing 1 of 2 buttons to receive an alcohol or water "drink" unit. Each alcohol "drink" targets a 7.5mg% increase in BrAC over 2.5 min. The water "drink" is an equal volume of saline.
Number of drinks per day | 10 days
  Participants will report the number of drinks they consume each day via EMA app added to their phone.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Weafer, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Northeastern University, Boston, Massachusetts
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No